CLINICAL TRIAL: NCT06860360
Title: The Face of Neuromuscular Dysfunction: Artificial Intelligence for the Analysis of Video Data of Facial Movement, with a Focus on Myasthenia Gravis
Brief Title: Artificial Intelligence for the Analysis of Video Data of Facial Movement, with a Focus on Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Delft University of Technology (Other)
Responsible Party: Principal Investigator, Martijn R. Tannemaat, MD PhD, MD PhD, Leiden University Medical Center
Other Study IDs: P20.083
Record Dates: First submitted 2022-08-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- myasthenia gravis
- healthy controls

SUMMARY:
Rationale: Myasthenia Gravis (MG) is an autoimmune disorder (AID) with antibodies against the NMJ, resulting in various degrees of muscle fatigability and weakness. All striated muscles can be involved, although the extra-ocular muscles are most commonly affected, giving rise to a fluctuating ptosis and diplopia. Facial muscles are also commonly affected, resulting in eye closure weakness, difficulty chewing and swallowing or speech impairments. Antibodies against the acetylcholine receptor (AChR) are present in over 80% of generalized MG patients. In the pure ocular form, AChR antibodies are detectable in nearly 50% of all patients. In approximately 4%, antibodies against the postsynaptic muscle-specific receptor tyrosine kinase (MuSK) are found and in 15% of the patients with generalized disease, no serum antibodies are detected1-3. Approximately 15% of AChR MG patients has a thymoma, in which case the disease can be classified as a paraneoplastic syndrome2. With a prevalence of 1 to 2 per 10.000, MG is considered a rare disease2.

The rarity of MG can make it difficult to diagnose, specifically for general Neurologists who are likely to encounter a patient with MG only a handful of times throughout their career. In addition, the fluctuating nature of the disease makes it difficult to make appropriate treatment decisions, especially as patients throughout the country are usually treated at one specialized center (in the Netherlands, the LUMC). Currently, patients who are in doubt whether they are experiencing an exacerbation have to make an appointment and travel for several hours to undergo assessment by their specialized Neurologist. An objective, reliable biomarker for disease severity that can be used at home would therefore greatly improve quality of life for many MG patients. Emerging possibilities in modern technologies can support doctors with all kinds of medical challenges, like offering diagnostic support, treatment decisions or patient follow-up. A technology of special interest for this study is advanced facial recognition. We aim to study the ability of existing software (FaceReader, Noldus) versus a deep learning model specifically developed for this purpose by the group of Jan van Gemert at the TU Delft to differentiate between healthy controls and patients with MG and between MG patients with different levels of disease severity.

Primary objectives:

To determine and compare the diagnostic yield of two different methods (FaceReader technology and a deep learning model specifically developed for video data) to analyse facial weakness from video recordings (04:00m) with different standardized facial expressions to:

1. Differentiate between MG patients and healthy controls.
2. Differentiate between mild and moderate to severe disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥ 18 years
* Subjects must understand the requirements of the study and provide written informed consent.

MG

* Clinical signs or symptoms suggestive of MG and at least one of the following:
* A serologic test for AChR antibodies or MuSK antibodies or
* A diagnostic electrophysiological investigation supportive of the diagnosis MG or
* A positive neostigmine test Healthy control group
* Volunteers from spouses, friends and family accompanying patient or employees from our department
* No medical conditions affecting the facial muscles, e.g. Graves' disease, previous stroke with a facial palsy
* No use of medication affecting the facial features, e.g. prednisone

Exclusion Criteria:

* Inability to give written informed consent
* Inability to read Dutch/ English video-instructions
* Participants with active Graves' disease or unilateral facial paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To answer the main objectives we will obtain a 04:00 min standardized facial video recording of MG patients in the outpatient clinic and Neurology ward, recorded at the LUMC. For the webcam recordings we will recruit participants from the Dutch-Belgian MG registry (P15.287). Informed consent forms of the MG registry with permission to be approached for future research are available.
  We will ask spouses and family to enrol as healthy controls, as well as employees of our department. The healthy control group will be age- and gender matched. Healthy controls are defined as subjects without medical conditions or medication which may influence the facial muscles, e.g. Graves thyroid disease, previous facial palsy due to a stroke or prednisone use. For the webcam recordings we will ask MG patients to introduce a healthy control of the same age.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
FaceReader | 2020-2023
  The primary parameter for the differentiation between healthy controls and MG and between different grades of MG disease severity with FaceReader is the diagnostic yield of individual muscles and combinations of muscles. The diagnostic yield is expressed as sensitivity, specificity and area under the curve of a receiver-operator curve (ROC) of the FaceReader algorithm. For this the quantitative data of facial weakness expressed in Action Units (AU), ranging between 0 (no activation) and +1 (maximal activation) will be used. Raw data from FaceReader provides the results of 20 AU's corresponding with 20 different facial movements of 20 facial muscles based on the Facial Action Coding System (FACS).
Narrow deep learning model | 2020-2023
  The primary parameter for the differentiation between healthy controls and MG and between different grades of MG disease severity with a working narrow deep learning model is the diagnostic yield. The diagnostic yield is expressed as sensitivity, specificity and area under the curve of a receiver-operator curve (ROC).
Disease severity | 2020-2023
  For comparison between different levels of disease severity the QMG score will serve as the gold standard. Groups based on disease severity are composed as following: mild QMG 0-9, moderate QMG 10-16 and severe QMG >16. For the home recording we will use the MG-Activities of Daily Living (MG-ADL) to measure disease severity since the QMG requires the physical presence of the patient. This is a commonly used tool in clinical trials. Groups based on disease severity are composed as following: mild MG-ADL 0-4, moderate-severe MG-ADL ≥5.

SECONDARY OUTCOMES:
Longitudinal changes | 2020-2023
  Detection of medication effects by obtaining multiple videos (longitudinal) in a subset of patients. The QMG score or MG-ADL is the parameter for change in disease severity. A previous study found a minimal clinically important difference (MCID) in QMG score of ≥2 for a baseline QMG score between 0 and 16. For a baseline QMG score >16 the MCID is ≥3 points change in QMG score4. For the MG-ADL the MCID is a change of ≥2 points5. For detection of medication effects, our aim is to detect an intra-participant change in QMG ≥2 or ≥3, depending of baseline QMG score. For the home recorded group our aim is to detect a change in MG-ADL score of ≥2 points.
FaceReader vs deep learning model | 2020-2023
  A comparison of the diagnostic yield of FaceReader parameters and classification by the deep learning model.
site versus home recording | 2020-2023
  A comparison of the diagnostic yield of FaceReader and the deep learning model of videos recorded in the standardized LUMC setting (green screen, lights, 4K camera) and home recorded videos using a webcam.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Tannemaat, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Raw data, including de-identified individual participants' data, that support the findings of this study are available from the corresponding author, upon reasonable request. Privacy laws preclude the sharing of facial videos of individual study participants.
Supporting Information: Study Protocol, SAP, ICF, CSR